CLINICAL TRIAL: NCT02928107
Title: Addressing Barriers to Adult Hearing Healthcare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Pro00070422; R21DC015003-01 (NIH); R33DC015003 (NIH); Pro00086182 (Other: Duke University Medical Center)
Record Dates: First submitted 2016-10-06; First posted 2016-10-10 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Hearing Loss; Geriatric Disorder
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- At-Home Telephone Screening (Tele-HS) (Experimental): Subjects receive printed educational materials about hearing loss and access to at-home Tele-HS
  Interventions: Other: Tele-HS
- PCP Encouragement, At-Home Tele-HS (Experimental): Subjects receives encouragement from primary care provider (PCP) or hearing screening, printed materials and access to at-home Tele-HS.
  Interventions: Other: Tele-HS; Other: PCP encouragement
- PCP Encouragement, In-Office Tele-HS (Experimental): Subjects receives PCP encouragement for hearing screening, printed materials and access to Tele-HS while in clinic.
  Interventions: Other: Tele-HS; Other: PCP encouragement
- CHEER Cohort (non-randomized) (No Intervention): Participants will complete a one page questionnaire related to Red Flag conditions during a routine Otolaryngology appointment for suspected hearing loss. The audiologist will be complete a questionnaire about the participants audiological assessment including Red Flag conditions. The Otolaryngology provider will complete a questionnaire about the participants otoscopic exam findings, Red Flag conditions, and indicate if any other conditions exist that me be considered a medical contraindication to hearing aid fitting.

INTERVENTIONS:
Other: Tele-HS — Patients will be given information on the Tele-HS and given access to take the screening at home or in-office, depending on arm.
  Arms: At-Home Telephone Screening (Tele-HS); PCP Encouragement, At-Home Tele-HS; PCP Encouragement, In-Office Tele-HS
Other: PCP encouragement — Patients will or will not either receive PCP encouragement to do the Tele-HS.
  Arms: PCP Encouragement, At-Home Tele-HS; PCP Encouragement, In-Office Tele-HS

SUMMARY:
The aim of this project is to develop evidence that can inform hearing health care best practices for adults between the ages of 65-75, and determine what level of involvement by the primary care practitioner (PCP) is required to inform and encourage adults age 65-75 to follow through with routine hearing screening.

This study also aims to evaluate the accuracy of assessment of medical conditions for which the FDA requires physician evaluation and management prior to hearing aid fitting, and determine which medical conditions should require medical evaluation prior to hearing aid fitting.

The results of this study should provide information to implement changes in health care policy to facilitate accessible and affordable hearing health care.

DETAILED DESCRIPTION:
Age-related hearing loss is the third-most common chronic condition affecting older adults in the US (data from Healthy People 2020 US Dept of Health and Human Services). This study aims to improve the understanding of attitudes, barriers and facilitators needed to improve hearing health care delivery. Two study cohorts of study participants between the ages of 65 - 75 are proposed.

The first cohort of participants include healthy adults being seen by a primary care provider (PCP) for a routine appointment. Each participating primary care practice is assigned to one of three different telephone hearing screening strategies that include progressive levels of PCP time and guidance to complete telephone-based hearing screening. Those who fail a telephone hearing screening go on to a medical referral study and receive (1) diagnostic audiological testing and (2) determination of the reliability and validity of identification of conditions that should require medical referral prior to hearing aid provision (called FDA 'Red Flag' conditions, including conditions such as sudden hearing loss, cerumen impaction, conductive hearing loss, dizziness, external deformity, ear drainage). We will evaluate the proportion of subjects in Groups 1 and 2 who dial the phone number and complete the telephone hearing test at or within two months of their PCP visit, relative to Group 3, and the proportion of subjects in all groups who: a) schedule and b) complete the visit for diagnostic audiological testing, and subsequently, c) complete a plan for appropriate hearing loss intervention, if indicated, within four months of initial hearing screening. Enrollment in this cohort is complete. 955 subjects were screened for eligibility. Of those, 660 patients were enrolled.

The second cohort includes adults who are being seen for a routine appointment for a complaint of hearing loss at one of several participating Ear, Nose, and Throat (ENT) practices in the CHEER network. Information about Red Flag conditions will be obtained from the patient, audiologist, and ENT provider. This information, along with Red Flag data from the PCP Cohort, will be used to evaluate the accuracy of assessment of medical conditions for which the FDA requires physician evaluation and management prior to hearing aid fitting, and determine which medical conditions should require medical evaluation prior to hearing aid fitting. Enrollment in this cohort is ongoing. The anticipated enrollment goal is 500 subjects.

ELIGIBILITY:
Primary Care Cohort:

Inclusion Criteria:

* 65-75 years of age
* Being seen by PCP for non-acute follow-up or annual appointment for primary care
* No prior history of hearing aid use or self-reported diagnosis of hearing loss

Exclusion Criteria:

* Not between the ages of 65-75
* Current or past hearing aid user
* Patient has been tested by an audiologist in the past and self-reports a hearing loss diagnosis
* Being seen by the PCP for an acute illness

CHEER Cohort:

Inclusion Criteria:

* 65-75 years of age
* Being seen by an OHNS/ENT provider for a complaint of hearing loss.
* Is scheduled to have an audiogram as standard of care for complaint of hearing loss.
* No prior diagnosis of hearing loss by a medical professional or history of hearing aid use

Exclusion Criteria:

* Not between the ages of 65-75
* Current or past hearing aid user
* Prior diagnosis of hearing loss or hearing aid user

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1146 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Completion of Tele-HS screen | 2 months of PCP appointment (day 1)
  The proportion (%) of subjects in Groups 1 and 2 who take the test will be compared to those in Group 3.
Medical conditions for which the FDA requires physician evaluation prior to hearing aid fitting | 1 day (following completion of Red Flag questionnaires by patient, audiologist and medical provider)
  Analysis of medical conditions for which the FDA requires physician evaluation prior to hearing aid fitting by comparing red flag assessments from patient, audiologist and ENT provider (CHEER Cohort)

SECONDARY OUTCOMES:
Scheduling of follow-up audiological testing | 4 months of date of Tele-HS
  The proportion (%) of subjects in Groups 1 and 2 who fail the Tele-HS and schedule follow-up testing compared to those in Group 3.
Completion of follow-up audiological testing | 4 months of date of Tele-HS
  The proportion (%) of subjects in Groups 1 and 2 who fail the Tele-HS and complete follow-up testing compared to those in Group 3.
Completion of plan for appropriate hearing loss intervention, if applicable | 4 months of date of Tele-HS
  The proportion (%) of subjects in Groups 1 and 2 who fail the Tele-HS, complete follow-up testing, and complete a plan for hearing loss intervention, if applicable, compared to those in Group 3.

OTHER OUTCOMES:
Significance of medical conditions requiring medical evaluation prior to hearing aid fitting | 1 day, completion of patient, audiologist and provider questionnaires
  Analysis to determine what medical conditions should require medical evaluation prior to hearing aid fitting (CHEER Cohort)
Cost to conduct telephone hearing screening in the Primary Care clinic setting | 1 day
  Cost to conduct hearing screening based on costs of educational material, telephone screening test, provider time and clinic space. (Both Cohorts)
Attitudes towards hearing loss | 2 days
  Analysis of attitudes towards hearing loss using the ALHQ questionnaire and focus group discussions
Attitudes of communication partners regarding hearing loss | 1 day, completion of the Significant Other Hearing Questionnaire (SOS-HEAR)
  Evaluation of how attitudes of significant others impact decision making to pursue hearing screening, diagnostic testing, and intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sherri Smith, PhD, Principal Investigator — Duke University
Locations (6):
- United States (6):
  - University of Michigan, Ann Arbor, Michigan
  - Northwell Health, New Hyde Park, New York
  - New York Eye and Ear of Mount Sinai, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Central Oregon ENT, Bend, Oregon
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
The data will be deposited into the Duke Research Data Repository (RDR), an openly accessible preservation archive maintained by the Duke University Libraries. The RDR will assign appropriate metadata (Dublin Core) for discoverability and provide a Digital Object Identifier (DOI) for persistent access and unique identification of the data. The data will be preserved in the RDR for the long-term according to RDR policies and procedures. When the data are transferred to the RDR, data curators will review deposits to help ensure they are complete and in a structure and format that supports long-term preservation, access, and reuse. The RDR provides for automated backup of all data, which provides an added layer of protection and security for the data.
Supporting Information: Study Protocol, SAP
Time Frame: At the end of the study data analysis

REFERENCES:
- [Derived] Dubno JR, Majumder P, Bettger JP, Dolor RJ, Eifert V, Francis HW, Pieper CF, Schulz KA, Silberberg M, Smith SL, Walker AR, Witsell DL, Tucci DL. A pragmatic clinical trial of hearing screening in primary care clinics: cost-effectiveness of hearing screening. Cost Eff Resour Alloc. 2022 Jun 25;20(1):26. doi: 10.1186/s12962-022-00360-5. PMID 35751122
- [Derived] Bettger JP, Dolor RJ, Witsell DL, Dubno JR, Pieper CF, Walker AR, Silberberg M, Schulz KA, Majumder P, Juhlin E, Smith SL, Francis HW, Tucci DL. Comparative implementation-effectiveness of three strategies to perform hearing screening among older adults in primary care clinics: study design and protocol. BMC Geriatr. 2020 May 11;20(1):170. doi: 10.1186/s12877-020-01576-x. PMID 32393184